CLINICAL TRIAL: NCT06090617
Title: The Water and Electrolytes Content in Salt-dependent Human HYpertension (WHYSKI) in the SKIn Before and After Surgical Cure of Primary Aldosteronism
Brief Title: Water and Electrolytes Content in HYpertension (WHYSKI) in the SKIn
Acronym: WHYSKI
Status: Recruiting | Type: Observational
Sponsor: University Hospital Padova (Other)
Responsible Party: Principal Investigator, Gian Paolo Rossi, MD, FAHA, FACC, Full Professor of Internal Medicine, MD, FAHA, FACC, University Hospital Padova
Other Study IDs: AOP1615
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Hyperaldosteronism; Hypertension; Aldosterone-producing Adenoma; Aldosteronism; Aldosterone Disorder; Essential Hypertension; Bilateral Adrenal Hyperplasia; Conn Adenoma
Keywords: Salt-dependent Hypertension; Primary Aldosteronism; Salt-sensitive; Blood Pressure; TonEBP; Tonicity Enhancing Binding Protein; RAAS; Renin Angiotensin Aldosterone System; BP; GAGs; Glycosaminoglycans
MeSH Terms: conditions — Hyperaldosteronism; Hypertension; Adrenocortical Adenoma; Essential Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- PA group 1: conclusive diagnosis of unilateral PA by the "four corners" criteria:
  1. Biochemical evidence of PA
  2. Lateralization of aldosterone secretion at adrenal venous sampling.
  3. Correction of biochemical values and fall of blood pressure after adrenalectomy.
  4. Immunohistochemical demonstration of CYP11B2 positive nodule(s)
  Interventions: Procedure: Skin Biopsy; Procedure: Video-laparoscopic adrenalectomy
- PA group 2: Presumed diagnosis of bilateral PA, defined as above but without evidence of lateralized aldosterone excess.
  Interventions: Procedure: Skin Biopsy
- PH Group: Primary (essential) Hypertension (PH): conclusively ascertained high blood pressure and exclusion of secondary hypertension
  Interventions: Procedure: Skin Biopsy
- Non Hypertensive Control Group: comprising patients submitted to surgery but free of hypertension
  Interventions: Procedure: Skin Biopsy

INTERVENTIONS:
Procedure: Skin Biopsy — Skin biopsies were obtained in all recruited patients.
Procedure: Video-laparoscopic adrenalectomy — Video-laparoscopic adrenalectomy in those with unilateral PA. (PA group 1)
  Groups: PA group 1

SUMMARY:
WHYSKI is a prospective within-patient observational clinical study designed to test the hypothesis that alterations of Na+, K+, water, and the lympho-angiogenetic transcription factor Tonicity Enhancing Binding Protein (TonEBP) mRNA take place in the interstitium of the skin compartment of patients with arterial hypertension due to primary aldosteronism in whom hypertension can be surgically cured.

DETAILED DESCRIPTION:
Background. Given the key role of Na+ in the pathophysiology of HT, this study will test the hypothesis that in PA, which is the paradigm of salt-dependent hypertension, the skin, Na+, K+ and water content is altered and these alterations are corrected by surgical cure of PA with video-laparoscopic adrenalectomy. The investigators will use skin biopsies to directly examine the content of Na+, K+, water, and the lympho-angiogenetic transcription factor Tonicity Enhancing Binding Protein (TonEBP) mRNA in the skin, an important reservoir of body Na+, in primary aldosteronism (PA), the prototype of salt-dependent hypertension.

Methods. The investigators will measure Na+, K+, and water content (by chemical-physical methods) and TonEBP mRNA copy number (by droplet digital PCR) in skin biopsies from a sex-mixed cohort of consecutive consenting patients with unilateral PA treated with a mineralocorticoid receptor antagonist (MRA), before surgery, at doses that correct hypokalemia and HT in order to refer them for surgery with normokalemia and controlled high blood pressure, as per protocol at our institution. The participants will be reassessed in an identical way again after surgical cure.

The investigators expect the dry weight (DW) of the skin specimen obtained at surgery to be significantly higher than at follow-up and to correlate positively with skin Na+, K+, and water content. Hence, if these predictions will be verified, the skin cations and water content will need to be DW-adjusted in order to provide meaningful comparisons across specimen obtained at different time points. The investigators expect the TonEBP mRNA copy number to be markedly overexpressed compared to healthy subjects.

The WHYSKI study will provide solid knowledge of the skin Na+, K+ and water content in patients with arterial salt-dependent hypertension due to PA, PH, and on the effect of cure of the hyperaldosteronism on these variables. The investigators also expect to gather novel knowledge on the molecular and cellular mechanisms involved in the regulation of the content on Na+, K+ and water in a compartment as the skin interstitium that has been largely neglected thus far.

ELIGIBILITY:
Inclusion Criteria:

PA Group

* Age: 18-75-year-old.
* Signed informed consent form.
* A diagnosis of PA defined as

  o Plasma aldosterone concentration > 15 ng/dL and aldosterone/renin ratio greater than 20.6 ng/mIU, measured after washout of interfering drugs or after changes of the drug treatment as previously detailed.
* Unilateral or bilateral evidence of PA at adrenal vein sampling

PH Group

* Age: from 18 to 75 years old
* Signed and dated informed consent form
* Diagnosis of essential hypertension defined either as:

  * Use of antihypertensive drug (s)
  * Arterial hypertension: in untreated patients this must be confirmed by daytime ambulatory blood pressure monitoring (ABPM), or home blood pressure monitoring, with blood pressure higher or equal to 135 mmHg for systolic blood pressure and/or higher or equal to 85 mmHg for diastolic blood pressure.
  * Exclusion of secondary hypertension by hormonal biochemical screening (aldosterone, renin, ARR<2.06 ng/dL:mIU/L, ACTH, 24h urine cortisol, morning plasma cortisol level, 24h urine metanephrines and catecholamines).

Control Group

* Age: from 18 to 75 years old
* Signed and dated informed consent form
* Normal arterial blood pressure defined either as:

  * None anti-hypertensive drug (s)
  * Normal arterial hypertension confirmed by daytime ambulatory blood pressure monitoring (ABPM), or home blood pressure monitoring, with blood pressure lower or equal to 135 mmHg for systolic blood pressure and/or lower or equal to 85 mmHg for diastolic blood pressure.
  * Exclusion of secondary hypertension by hormonal biochemical screening (aldosterone, renin, ACTH, 24h urine cortisol, morning plasma cortisol level, 24h urine metanephrines and catecholamines).

Exclusion Criteria:

PA Group

* history of allergy/intolerance to local anesthesia;
* refusal of the patient to undergo skin biopsy;
* refusal of the patient to undergo AVS, and/or contraindications to the general anesthesia that is required for laparoscopic adrenalectomy and/or to undergo adrenalectomy if indicated;
* cortisol-aldosterone co-secreting adenoma or pheochromocytoma. PH Group and Control Group
* Concurrent skin diseases, for example psoriasis, and any pathological conditions that, in the judgement of the investigators, could affect skin electrolyte and water content.
* Subjects with diabetes mellitus type 1 and 2, as drugs affecting the renin-angiotensin-aldosterone system and/or renal Na+ handling as, for example, SGLT-2 inhibitors (gliflozins) 16 were considered to potentially bias results.
* Other conditions characterized by possible lymphatic disruption such as lipedema, cyclic idiopathic edema, lymphedema, and malignancies were also exclusion criteria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients referred to either the Endocrine Surgery unit, the Specialized Center for Blood Pressure Disorders of Regione Veneto of the Azienda Ospedale-Università di Padova, or other surgery departments of the same institution were recruited.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
measure the Na+, K+ and water content in the skin of patients with primary aldosteronism (PA, PA Group), primary (essential) hypertension HT patients (PH Group) and in normotensive patients (Control Group). | Baseline (Surgery), Month 1 after Surgery (for PA Group 1 only)
  With validated chemical physical methods, we will measure the Na+, K+ and water content in the skin of patients with primary aldosteronism (PA, PA Group), primary (essential) hypertension HT patients (PH Group) and in normotensive patients (Control Group). The skin biopsy will be performed during adrenalectomy in consecutive patients with confirmed unilateral PA (PA Group) and in parallel in the same anatomical region in the PH group and in the Control Group, during surgery for benign diseases.
  To verify if the cure of PA improves Na+, K+ and water skin clearance in the PA Group the skin biopsy obtained during adrenalectomy will be within-patient compared to that obtained one month after adrenalectomy (PA Group 1). In PA patients found not to have unilateral PA (PA Group 2), the biopsy will be obtained after one month of target medical treatment with canrenone, a mineralocorticoid receptor antagonist.

SECONDARY OUTCOMES:
mRNA content of Tonicity-Enhancing Binding Protein TonEBP (also known as NFAT5) | Baseline (Surgery), Month 1 after Surgery (for PA Group 1 only)
  While the measurement of skin Na+, K+ and water is the main study outcome, an additional important goal will be to determine the molecular mechanisms driven by "skin sodium storage" that underlie the crosstalk between skin cells, macrophages and lymphatic vessels in the interstitium of the patient with PA (PA group 1) and essential hypertensive patients (EH Group) compared with the normotensive patient (Control Group). To this end we will explore the mRNA content of Tonicity-Enhancing Binding Protein TonEBP (also known as NFAT5), a transcription factor known to activate neo-lymphoangiogenesis, using molecular biology techniques.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedale Università di Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: Yes
IPD available on reasonable request but if consistent with the ongoing privacy legislation.

REFERENCES:
- [Background] Wiig H, Luft FC, Titze JM. The interstitium conducts extrarenal storage of sodium and represents a third compartment essential for extracellular volume and blood pressure homeostasis. Acta Physiol (Oxf). 2018 Mar;222(3). doi: 10.1111/apha.13006. Epub 2017 Dec 20. PMID 29193764
- [Background] Rossier BC, Bochud M, Devuyst O. The Hypertension Pandemic: An Evolutionary Perspective. Physiology (Bethesda). 2017 Mar;32(2):112-125. doi: 10.1152/physiol.00026.2016. PMID 28202622
- [Background] Rossi GP, Bisogni V, Bacca AV, Belfiore A, Cesari M, Concistre A, Del Pinto R, Fabris B, Fallo F, Fava C, Ferri C, Giacchetti G, Grassi G, Letizia C, Maccario M, Mallamaci F, Maiolino G, Manfellotto D, Minuz P, Monticone S, Morganti A, Muiesan ML, Mulatero P, Negro A, Parati G, Pengo MF, Petramala L, Pizzolo F, Rizzoni D, Rossitto G, Veglio F, Seccia TM. The 2020 Italian Society of Arterial Hypertension (SIIA) practical guidelines for the management of primary aldosteronism. Int J Cardiol Hypertens. 2020 Apr 15;5:100029. doi: 10.1016/j.ijchy.2020.100029. eCollection 2020 Jun. PMID 33447758
- [Background] Elijovich F, Weinberger MH, Anderson CA, Appel LJ, Bursztyn M, Cook NR, Dart RA, Newton-Cheh CH, Sacks FM, Laffer CL; American Heart Association Professional and Public Education Committee of the Council on Hypertension; Council on Functional Genomics and Translational Biology; and Stroke Council. Salt Sensitivity of Blood Pressure: A Scientific Statement From the American Heart Association. Hypertension. 2016 Sep;68(3):e7-e46. doi: 10.1161/HYP.0000000000000047. Epub 2016 Jul 21. No abstract available. PMID 27443572
- [Derived] Torresan F, Rossi FB, Caputo I, Zanin S, Caroccia B, Mattarei A, Paccagnella M, Kohlscheen E, Seccia TM, Iacobone M, Rossi GP. Water and Electrolyte Content in Hypertension in the Skin (WHYSKI) in Primary Aldosteronism. Hypertension. 2024 Dec;81(12):2468-2478. doi: 10.1161/HYPERTENSIONAHA.124.23700. Epub 2024 Oct 2. PMID 39355924
- [Derived] Torresan F, Rossi FB, Zanin S, Caputo I, Caroccia B, Iacobone M, Rossi GP. Water and Electrolyte Content in Salt-Dependent HYpertension in the SKIn (WHYSKI): Effect of Surgical Cure of Primary Aldosteronism. High Blood Press Cardiovasc Prev. 2024 Jan;31(1):15-21. doi: 10.1007/s40292-023-00614-0. Epub 2023 Dec 21. PMID 38123759